CLINICAL TRIAL: NCT05338398
Title: A Phase 1/Phase 2 Study for the Prevention of Oral Mucositis (SPOM)
Brief Title: Study for the Prevention of Oral Mucositis (SPOM)
Acronym: SPOM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: E2Bio Life Sciences, LLC (Industry)
Collaborators: Hematology Center after Prof. R. Yeolyan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BL002
Record Dates: First submitted 2022-04-11; First posted 2022-04-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Chemotherapy; Inflammation; Benzydamine; Bocaliner; Medical Device; Prevention; Intervention; Pain; Oral Ulcerations
MeSH Terms: conditions — Stomatitis; Inflammation; Pain; Oral Ulcer | interventions — Benzydamine; Anti-Inflammatory Agents

STUDY DESIGN:
Intervention Model Description: Control Group (Group 1):
  Standard Therapy Hematologic malignancy Saline mouthwash (±Bocaliner™)
  Intervention Group (Group 2):
  Benzydamine mouthwash Hematologic malignancy Benzydamine mouthwash (±Bocaliner™)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (Group 1): Standard Therapy (Placebo Comparator): Group 1 will receive standard therapy with conventional oral care to prevent oral mucositis consisting of oral hygiene and rinses/mouthwashes with saline solutions 3-5 times daily.
  Half of the subjects in Group 1 will also receive Bocaliner™ devices
  Interventions: Device: Bocaliner
- Intervention Group (Group 2): Benzydamine mouthwash (Experimental): Group 2 will receive benzydamine mouthwashes 3-5 times daily. Half of the subjects in Group 1 will also receive Bocaliner™ devices.
  Interventions: Drug: Benzydamine

INTERVENTIONS:
Device: Bocaliner — Bocaliner is a soft, orally inserted device that has been demonstrated to increase the oral retention of oral, topical therapies such as mouthwashes and gels.
  Other Names: Oral topical medication retention device
  Arms: Control Group (Group 1): Standard Therapy
Drug: Benzydamine — Benzydamine is an anti-inflammatory and antibiotic mouthwash that has shown promise for the treatment of radiation-induced oral mucositis.
  Other Names: Anti-inflammatory and antibiotic mouthwash
  Arms: Intervention Group (Group 2): Benzydamine mouthwash

SUMMARY:
1. Study Design

   * Prospective, Randomized, Questionnaire-Based Study
   * Study Type: Phase 1/Phase 2 Interventional Clinical Trial
   * Intervention Model: Parallel Assignment
   * Masking: None (Open-label)
   * Actual Enrollment: 100 participants
   * Allocation: Randomized
   * Primary Purpose: Supportive Care/Treatment
   * Study groups
   * Control Group (Group 1): Saline mouthwash (±Bocaliner™)
   * Intervention Group (Group 2): Benzydamine mouthwash (±Bocaliner™)
2. Settings

   * Single-center (a specialized hematology center)
   * Location: Hematology Center after Prof. R. Yeolyan, 7 Nersisyan St, Yerevan 0014, Armenia
   * Subjects will initially be enrolled, consented, examined, and complete initial questionnaires in the healthcare provider's office Subjects will undergo initial evaluation and follow-up examinations to determine WHO Oral Mucositis Scores
   * Subjects will complete questionnaires at the medical center with the Research Coordinator 7 and 14 days after study enrollment. Subjects using Bocaliner™ will additionally complete a follow-up questionnaire.
   * Application of Bocaliner™ will be carried out first at the hospital followed by self-administration at home.

DETAILED DESCRIPTION:
This is a single-center randomized controlled trial . The goal of this study is to find whether topical benzydamine is superior in preventing chemotherapy-induced oral mucositis compared to standard methods, which include oral rinses with saline. This study also aims to determine the tolerance and response to the use of Bocaliner™ (a new medical device designed to improve treatment and prevention of oral mucositis) in the prevention of oral mucositis.

All patients will be referred by their treating physicians to the designated study healthcare providers. Patients undergoing chemotherapeutic treatment for a diagnosed hematologic malignancy and at risk for oral mucositis will be enrolled. All subjects will sign an informed consent form prior to enrollment.

Initially, subjects will undergo a general oral examination to determine any significant dental or oral problems. Patients will be examined by study team members for potential eligibility. Subjects will then be randomized into two groups. Group 1 will receive standard therapy with conventional oral care to prevent oral mucositis consisting of oral hygiene and rinses/mouthwashes with saline solutions 3-5 times daily for at least 2 consecutive weeks. Group 2 will receive benzydamine mouthwashes 3-5 times daily for at least 2 consecutive weeks. Half of the subjects in each group will also receive Bocaliner™ devices along with cleaning materials with instructions about device use and cleaning based on another randomization. Bocaliner™ will be used with each topical treatment (either standard treatment or benzydamine mouthwash) for oral mucositis 3-5 times per day for 2 weeks. Allocation to each study group as well as the receipt of Bocaliner™ as an adjunct to the prevention strategy will be determined by randomization.

Subjects assigned to receive Bocaliner™ will initially place the device inside of their mouth for 5 minutes and fill out the Initial Bocaliner™ Questionnaire. The subjects will then continue all original therapy for oral mucositis including oral topical treatments and will place the Bocaliner™ device inside of their mouth and hold it in place up to 40 minutes as instructed after each topical treatment. The device is hypothesized to improve the effects of treatments.

All subjects will be contacted by the Research Coordinator at 7 and 14 days after enrollment and undergo an oral examination using the WHO Oral Toxicity Scale (Days 7 and 14). Subjects receiving Bocaliner™ will describe their use of the device on the Bocaliner™ Follow up Questionnaire (Day 14). Subjects are instructed to contact their physicians whenever oral mucositis develops. Following detailed examination, the subjects will be asked to answer the questions from the Modified PROMS Questionnaire.

Objectives A.To determine the initial level of tolerance to the placement inside of their mouth and the use of Bocaliner™ in subjects undergoing chemotherapy B.To collect patient-reported effects of the use of Bocaliner™ in combination with oral topical medications for the prevention of oral mucositis.

C. To determine the efficacy of benzydamine mouthwash in the prevention of oral mucositis in patients undergoing chemotherapy for hematologic malignancies D. To determine the efficacy of Bocaliner™ addition in enhancing the preventive effects of different mouthwashes.

1. BACKGROUND/LITERATURE REVIEW Oral mucositis, defined as an inflammation of the mucosal lining of the mouth causing redness, soreness, and mouth pain, is a serious complication of cancer treatment involving chemotherapy and/or radiotherapy. In some cases, the pain becomes so severe that patients cannot eat or keep up with fluid intake. Management of these patients often requires the prescription of opioid pain medications and further hospitalization for advanced nutritional and supportive therapy. Oral mucositis negatively impacts the quality of life in patients receiving cancer treatment. When severe, oral mucositis may require patients to delay or discontinue their treatment for cancer.

Oral mucositis occurs in 20-40% of all patients receiving chemotherapy and in 80% of patients receiving stem cell transplantation. The Multinational Association for Supportive Care in Cancer (MASCC) has developed guidelines for preventing and treating oral mucositis, providing recommendations regarding different groups of interventions. Preventive measures that may be effective include basic oral care, anti-inflammatory agents, intraoral photobiomodulation, cryotherapy, growth factors, and natural agents.

Several products aiming at reducing oral mucositis rates in patients undergoing cancer treatment were proposed, including various types of mouthwash, gels, and rinses. Preparations recommended for use in the treatment of oral mucositis may contain morphine or doxepin. Lidocaine, either alone or combined with diphenhydramine, saline, sodium bicarbonate, and magnesium/aluminum hydroxide is also used. Another group of products is applied to protect the mucosal surfaces of the oral cavity (mucosal-protective agents); however, the evidence regarding the efficacy of these agents has been limited. The current guidelines by MASCC do not have specific recommendations regarding the use of these topical agents, other than morphine mouthwash for pain.

Preparations recommended by the expert panel for the prevention of OM include oral glutamine, intravenous KGF-1, intraoral photobiomodulation, honey, and benzydamine mouthwash. These recommendations, however, are given to specific patient populations, such as those undergoing autologous hematopoietic stem-cell transplantation or individuals with head and neck cancer undergoing radiotherapy or combined radio-chemotherapy.

Oral topical applications (e.g., gels, rinses, and mouthwashes) are usually swished in the mouth and then spit out, thus remaining inside the oral cavity from 10 seconds up to minutes only. This brief period inside the mouth likely limits their healing or analgesic effects on the oral mucosa. The efficacy of topical treatments largely depends on the ability of an agent to stick to the mucosa. The removal of these medications is facilitated by dilution by the saliva, constant muscular movements, and ongoing swallowing. The combined effects of these factors are thought to further limit the efficacy of different agents on the oral mucosa.

Bocaliner™ is a soft and lightweight medical device that has been scientifically engineered to help patients with oral mucositis. The device is constructed from silicone rubber that is designed to be worn comfortably by patients while the subjects are using mouthwashes and gels to prevent or treat oral mucositis. Bocaliner™ effectively prolongs the time of a topical polymer remaining inside the oral cavity and increases the area under the curve of the polymer versus the time curve. Bocaliner™ is hypothesized to keep topical treatments in the mouth longer by covering a larger surface of the oral mucosa, reducing salivary dilution, and holding the mouth still after the application of oral topical therapies. These effects are hypothesized to prolong the protective or healing effects of various agents and thus improve the prevention or treatment of oral mucositis.

1. Population Adult patients undergoing chemotherapy for hematologic malignancies and at risk for the development of oral mucositis.
2. Sample Size The study plans to enroll 88 patients. A power calculation was performed. Based on the currently available literature, it is anticipated that 35% of subjects in Group 1 will develop oral mucositis and 10% of subjects in Group 2 will develop oral mucositis. For alpha of 0.05 and 80% power, the investigators will need 44 subjects in each group, making it a total of 88 participants.
3. Recruitment Healthcare providers including oncologists and oncology nurses, specializing in the care of patients with hematologic malignancies will be referral sources for the study.
4. Study Procedures

   1. Patient Inclusion
   2. Randomization into 2 study groups
   3. Tryout and initial assessment of Bocaliner™ in assigned patients
   4. Treatment with topical oral agents for prevention of oral mucositis
   5. Collection of patient-reported outcomes and follow-up assessment
   6. Follow-up evaluation of Bocaliner™ in assigned patients at 14 days
5. Randomization Block randomization will be used with two strata: sex and use of Bocaliner™. Each block will be initially randomized to either a control treatment with saline rinses or an investigational treatment with benzydamine oral mouthwash. Each block will consist of 4 subjects with a 1:1 allocation of men and women. The subjects will further be randomized to receive treatment adjunct with the Bocaliner™ device or not. The decision to receive rinses with saline will be defined according to the preferences of each patient and their treating physicians.

   2. DATA MANAGEMENT PLAN All electronic records containing patient data will be stored in a password-protected electronic data file on a password-protected computer. Similarly, all paper files and printed documents will be stored in a locked file cabinet with key access only available to the principal investigator and study coordinator. The sponsoring organization will receive de-identified file(s) with randomly assigned numbers (e.g., 1-75) instead of patients' names or initials.

   3. DATA COLLECTION Upon receiving informed consent, the demographic data from each participant will be collected during the first visit by research assistants using case report forms

   4. DATA ANALYSIS Phase 1 tolerability and safety data for the Bocaliner™ device will be assembled in tabular form and analyzed separately. Data for subjects in Group 1 and Group 2 will be assembled in tabular form. Oral mucositis incidences, pain scores, and total scores between Group 1 and Group 2 from the questionnaires will be compared using nonparametric statistical tests. A comparison of the percentage of patients that achieve the primary endpoint between the two groups will be performed using cross-table analysis. Multivariate analysis will be used to identify measured parameters that are associated with improvement in oral mucositis.

   5. BENEFITS Benzydamine mouthwash has been studied and recently recommended for the prevention of oral mucositis in patients with head and neck cancer undergoing moderate-dose radiotherapy or suggested for those who receive combined radiotherapy-chemotherapy treatment. The benefits of this mouthwash in chemotherapy patients have not been determined.

   Enrolled subjects additionally receiving Bocaliner™ (as an adjunct to saline rinses or benzydamine mouthwash) may experience a clinical improvement or prevention of oral mucositis, a condition that has few treatment options at this time but has a detrimental impact on the life of affected patients. All study subjects will receive a $20 gift card upon completion of the study.

   6. RISKS Bocaliner™ is registered with the Food and Drug Administration (FDA) as a Class I Medical Device. This designation suggests that Bocaliner™ has a very low risk for adverse events.

   Benzydamine is known to be a well-tolerated topical medication. In some individuals, numbness or a sense of stinging, burning, and itching may happen. Other rare risks may include skin rash, nausea, diarrhea, swelling, or cough.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed hematologic malignancy
* Ongoing chemotherapeutic treatment
* Properly obtained written informed consent
* Age of 18 years or older
* Willingness to use the study materials for at least 2 weeks, including

  * Bocaliner™ device
  * Benzydamine mouthwash
  * Saline or baking soda mouthwash

Exclusion Criteria:

* No informed consent
* Systemic disease affecting oral mucosa
* Recurrent oral lesions other than oral mucositis
* Age of less than 18 years
* Recent invasive procedures of the mouth
* Use of medications affecting salivation (cholinergic, cholinomimetic, anti-cholinergic)
* Concurrent or previous radiotherapy
* Oral or maxillofacial disorders
* Inability/unwillingness to wear Bocaliner™ for the study period
* Unwillingness to use mouthwashes
* Known intolerance to silicone materials
* Known intolerance to benzydamine or any component of the formulation
* Individuals with significant difficulties to communicate and understand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis Incidence (WHO Oral Toxicity Scale) during 2 weeks of follow-up | Week 2
  A standard evaluation based on physical appearance of the oral mucosa and history

SECONDARY OUTCOMES:
Change in Modified Patient-Reported Oral mucositis Symptom Score by 30 percent at 7 and 14 days. (Minimum Score 0, Maximum Score 1200). Higher Scores Mean Worse Outcome. | Week 1 and 2
  Patient reported outcome related to severity of symptoms and effect of oral mucositis
Severity of oral mucositis (changes in World Health Organization's Oral Toxicity Scale). Minimum grade = 0, maximum grade= 4. Higher grade indicates worse outcome. | Week 1 and 2
  A standard evaluation based on physical appearance of the oral mucosa and history
Duration of oral mucositis (documented by the treating physician) | Week 3
  A clinical determination by the treating physician
Pain associated with oral mucositis (Modified Patient-Reported Oral mucositis Symptoms Score). Minimum score = 0, maximum score= 100. Higher score indicates worse outcome. | Week 1 and 2
  Patient reported outcome related to severity of pain

OTHER OUTCOMES:
Safety and Tolerability of Bocaliner, an Orally Inserted Device in Patients Undergoing Chemotherapy (Phase 1 Trial) | Baseline and week 2. (No score utilized. Descriptive analysis only.). Phase 1 data will be analyzed separately
  Patient reported outcome from questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Yervand Hakobyan, MD, Principal Investigator — Hematology Center after Prof. R. Yeolyan
Locations (1):
- Hematology Center after Prof. R. Yeolyan, Yerevan, Armenia

REFERENCES:
- [Background] Daugelaite G, Uzkuraityte K, Jagelaviciene E, Filipauskas A. Prevention and Treatment of Chemotherapy and Radiotherapy Induced Oral Mucositis. Medicina (Kaunas). 2019 Jan 22;55(2):25. doi: 10.3390/medicina55020025. PMID 30678228
- [Background] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Background] Elad S, Yarom N. The Search for an Effective Therapy and Pain Relief for Oral Mucositis. JAMA. 2019 Apr 16;321(15):1459-1461. doi: 10.1001/jama.2019.3269. No abstract available. PMID 30990535
- [Background] Sio TT, Le-Rademacher JG, Leenstra JL, Loprinzi CL, Rine G, Curtis A, Singh AK, Martenson JA Jr, Novotny PJ, Tan AD, Qin R, Ko SJ, Reiter PL, Miller RC. Effect of Doxepin Mouthwash or Diphenhydramine-Lidocaine-Antacid Mouthwash vs Placebo on Radiotherapy-Related Oral Mucositis Pain: The Alliance A221304 Randomized Clinical Trial. JAMA. 2019 Apr 16;321(15):1481-1490. doi: 10.1001/jama.2019.3504. PMID 30990550
- [Background] Kushner JA, Lawrence HP, Shoval I, Kiss TL, Devins GM, Lee L, Tenenbaum HC. Development and validation of a Patient-Reported Oral Mucositis Symptom (PROMS) scale. J Can Dent Assoc. 2008 Feb;74(1):59. PMID 18298885
- [Background] Abstracts for MASCC/ISOO Annual Meeting 2019. Support Care Cancer. 2019 May 18:1-302. doi: 10.1007/s00520-019-04813-1. Online ahead of print. No abstract available. PMID 31102057
- [Background] Jones JA, Avritscher EB, Cooksley CD, Michelet M, Bekele BN, Elting LS. Epidemiology of treatment-associated mucosal injury after treatment with newer regimens for lymphoma, breast, lung, or colorectal cancer. Support Care Cancer. 2006 Jun;14(6):505-15. doi: 10.1007/s00520-006-0055-4. Epub 2006 Apr 7. PMID 16601950
- [Background] Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, McGuire DB, Migliorati C, Nicolatou-Galitis O, Peterson DE, Raber-Durlacher JE, Sonis ST, Elad S; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2014 May 15;120(10):1453-61. doi: 10.1002/cncr.28592. Epub 2014 Feb 25. PMID 24615748
- [Background] Vera-Llonch M, Oster G, Ford CM, Lu J, Sonis S. Oral mucositis and outcomes of allogeneic hematopoietic stem-cell transplantation in patients with hematologic malignancies. Support Care Cancer. 2007 May;15(5):491-6. doi: 10.1007/s00520-006-0176-9. Epub 2006 Dec 1. PMID 17139495
- [Derived] Oganesyan A, Harutyunyan L, Vanoyan A, Martirosyan N, Badikyan M, Gregory M, Oganesyan T, Ghahramanyan N, Ehrenpreis ED, Hakobyan Y. Tolerability and safety of a new oral device for prevention and treatment of oral mucositis in patients with hematologic malignancies undergoing chemotherapy. Support Care Cancer. 2025 Jul 31;33(8):733. doi: 10.1007/s00520-025-09722-0. PMID 40742572